CLINICAL TRIAL: NCT04870801
Title: Evaluation of Respirogen Oxygen Microbubble Technology: Efficacy for Human Use During Rest in Normal and Low-oxygen Environments
Brief Title: An Alternative Way To Deliver Oxygen To People
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The project was denied funding and the protocol was subsequently closed. No participants were enrolled.
Sponsor: Christopher Bell (Other)
Collaborators: Respirogen Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-10219H
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Following screening, six healthy adults will report to the Human Performance Clinical Research Laboratory on two separate occasions, each separated by ~7-14 days. During each visit, study participants will undergo physiological monitoring prior to and during inhalation of hypoxic (FiO2=0.15) gas mixtures. During one of these visits, following initiation of hypoxic gas breathing, colon administration of RMO will commence.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Oxygen Visits without Respirogen Micro-Oxygen (No Intervention): During each visit, study participants will undergo physiological monitoring prior to and during inhalation of hypoxic (FiO2=0.15) gas mixtures.
- Low Oxygen Visits with Respirogen Micro-Oxygen (Experimental): During each visit, study participants will undergo physiological monitoring prior to and during inhalation of hypoxic (FiO2=0.15) gas mixtures.
  Interventions: Drug: Respirogen Micro-Oxygen

INTERVENTIONS:
Drug: Respirogen Micro-Oxygen — Enteral (rectal) delivery of Respirogen Micro-Oxygen
  Arms: Low Oxygen Visits with Respirogen Micro-Oxygen

SUMMARY:
The availability of oxygen is a crucial prognostic indicator for outcomes pertinent to many chronic diseases. Accordingly, interventions that might increase oxygen availability have obvious beneficial clinical application. In this regard, Respirogen Micro-Oxygen (RMO) technology holds considerable promise. Data from experimental animal models of lung injury suggest administration of RMO is a feasible method to deliver oxygen in a manner independent of pulmonary function. Our ultimate long-term goal is to provide a product that can be used to deliver oxygen to humans experiencing respiratory distress and pulmonary dysfunction In this first exploratory study, our goal is to begin to understand the physiological responses to enteral (rectal) delivery of RMO in low-oxygen environments in healthy adults at rest.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-40 years,
* body mass index between 19 and 30 kg/m^2,
* resident at a similar altitude for a minimum of 1-year,
* no travel to/from areas varying by ~2000 feet of elevation within 4-weeks of initiation of study participation.

Exclusion Criteria:

* identification of overt chronic disease (including cardio-pulmonary disorders),
* prior diagnosis of asthma, cystic fibrosis, Chronic obstructive pulmonary disease, or ventilator therapy
* anemia,
* pregnancy,
* habitual use of tobacco/nicotine products,
* known allergy to sodium phosphate (or other common laxatives),
* habitual use of recreational drugs that require inhalation,
* history of seizures, kidney problems, stomach or bowel problems, ulcerative colitis, problems with swallowing or gastric reflux, gout, and and/or low blood sodium.
* irritable bowel
* ACUTE respiratory illness such as bronchitis, pneumonia, Upper Respiratory Infection OR ACUTE GI issues such as gastroenteritis.
* Anemia (as measurement of hemoglobin and/or hematocrit) .
* sickle cell disease.
* history of altitude sickness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Increases Oxygen saturation (SpO2) with RMO | Randomized crossover, visits separated by a minimum 7 days and maxim 14 days
  Enteral (rectal) delivery of without and with RMO to resting adult men and women during short-term breathing of hypoxic gas mixtures.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Bell, PhD, Principal Investigator — CSU
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No